CLINICAL TRIAL: NCT00269464
Title: Chronic Schizophrenia With Obsessive-Compulsive Symptoms: Comorbidity or a Subtype?
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-03-8888-JZ-CTIL
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia; Obsessive Compulsive Disorder
MeSH Terms: conditions — Schizophrenia; Obsessive-Compulsive Disorder

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Evaluating the prevalence and characteristics of obsessive-compulsive (OC) symptoms in patients with chronic schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic patients
* Schizophrenic patients with OCD

Exclusion Criteria:

* Organic problems

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University